CLINICAL TRIAL: NCT04725786
Title: Pertinence Clinique de l'échographie Thoracique Pour le Diagnostic précoce de la Pneumopathie Interstitielle Diffuse de la sclérodermie systémique - Etude Pilote
Brief Title: Clinical Relevance of Thoracic Echography for the Early Diagnosis of Interstitial Lung Disease in Systemic Scleroderma - Pilot Study
Acronym: PRECOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DR20098; 2020-A03249-30 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2021-01-13; First posted 2021-01-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2022-06

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case group (Experimental): The intervention of the research corresponds to the realization of a thoracic echography.
  Interventions: Other: thoracic echography

INTERVENTIONS:
Other: thoracic echography — The research intervention corresponds to the performance of a thoracic echography to diagnose an incipient pulmonary interstitial syndrome.

SUMMARY:
Diffuse interstitial lung disease (PID) is the leading cause of death in systemic scleroderma (SSc). Major progress has recently been made in its therapeutic management. Early diagnosis is essential to optimize this management. Current diagnostic techniques are based on high-resolution computed tomography on the thorax (HRCT) and pulmonary functional tests (PFT). However, these explorations have their limitations. Thus, there is a need for new techniques for a very early diagnosis of PID-SSc.

Thoracic ultrasound (TUS) is an innovative, easily accessible, non-irradiating, inexpensive and painless tool. It is an emerging technique for the diagnosis of PID and has already proven its sensitivity for the detection of interstitial damage, as defined by HRCT.

The main objective of the PRECOSS study is to describe the prevalence of an ultrasound interstitial syndrome in patients with SSc, free of PID-SSc (defined by the Goh criteria) detectable by HRCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of systemic scleroderma according to EULAR/ACR 2013 criteria
* Absence of diffuse interstitial lung disease proven by scanner on the day of inclusion
* Forced vital capacity ≥ 80% of the value predicted on the last respiratory function test performed.
* Carbon monoxide diffusion capacity corrected for hemoglobinemia ≥ 70% of the value predicted on the last respiratory function test performed.
* Patient capable of performing functional exploration during the year
* Affiliation to a social security system
* Patient who has given free and informed consent

Exclusion Criteria:

* Any other connectivity associated to systemic sleroderma
* Any chronic pathologies, co-morbidities, history judged by the investigator as being likely to lead to complications for the patient and/or which may impact the results of functional exploration during exercise.
* All known fibrotic and/or obstructive respiratory pathologies.
* Presence of echocardiographic signs of pulmonary arterial hypertension according to 2015 criteria
* Diagnosis of left heart disease
* Cumulative smoking > 10 packs.years
* Infectious pneumonia within 90 days prior to inclusion
* Acute respiratory illness requiring hospitalization within one year prior to inclusion
* Pregnant or breastfeeding woman
* Refusal to participate in the study
* Refusal to use the data
* Adults under legal protection (temporary protection measure, curatorship, guardianship)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Presence of interstitial syndrome on echography | At baseline
  Interstitial syndrome is defined by the total number of B lines is greather than or equal to 10 and/or the average thickness of the pleural line is greater than 3 mm on at least one test site and/or the irregularity score of the pleural line is greater than 16%

SECONDARY OUTCOMES:
Ventilatory mechanics | At Baseline
  Measured by spirometry
Ventilatory mechanics | At Baseline
  Measured by plethysmography
Ventilatory mechanics | At Baseline
  Measured by impulse oscillometry
Ventilatory mechanics | At Baseline
  Measured by cardiopulmonary exercise testing
Pulmonary gas exchange | At Baseline
  Measured by cardiopulmonary exercise testing
Pulmonary gas exchange | At baseline
  Measured by Diffusing capacity for carbon monoxide
Pulmonary gas exchange | At baseline
  Measured by 6-minute walk test
Exercise capacity | At baseline
  Measured by cardiopulmonary exercise testing
Circulatory response | At baseline
  Measured by cardiopulmonary exercise testing
Dyspnoea | At baseline
  Measured by cardiopulmonary exercise testing
Dyspnoea | At baseline
  Assessed by Dyspnea12
Dyspnoea | At baseline
  Assessed by Modified Medical Research Council (mMRC) Scale
Assessment of Quality of life | At baseline
  Assessed by Cochin 17-item Scleroderma Functional Scale
Assessment of Quality of life | At baseline
  Assessed by Saint George's Respiratory Questionnaire (SGRQ)
Cough | At baseline
  Evaluation by Leicester Cough Questionnaire - French translation

OTHER OUTCOMES:
Nailfold capillaroscopy | At baseline
  Classification of Cutulo

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Tours, Tours, France

REFERENCES:
- [Result] Mercier C, Thoreau B, Flament T, Legue S, Pearson A, Jobard S, Marchand-Adam S, Plantier L, Diot E. High Prevalence of the Lung Ultrasound Interstitial Syndrome in Systemic Sclerosis Patients with Normal HRCT and Lung Function-A Pilot Study. J Clin Med. 2024 May 14;13(10):2885. doi: 10.3390/jcm13102885. PMID 38792426